CLINICAL TRIAL: NCT01924780
Title: Evaluation of the Anti-inflammatory Potential of NEMOS® Transcutaneous Vagus Nerve Stimulation Device in Patients With Juvenile Idiopathic Arthritis
Brief Title: NEMOS in Normal Volunteer and JIA Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karin Palmblad (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Karin Palmblad, M.D. PhD Senior scientist, Astrid Lindgren Children´s Hospital
Organization: Astrid Lindgren Children´s Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEMOS1
Record Dates: First submitted 2013-08-12; First posted 2013-08-16 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Inflammatory Response
Keywords: Dose-Response Relationship, Immunologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NEMOS device stimulation 10 minutes (Active Comparator): Subject will be stimulated in the cymba concha with a vibro-tactile mechanical device for 10 minutes
  Interventions: Device: Stimulation 10 minutes; Device: NEMOS transvagal stimulation 60 minutes; Device: NEMOS Device sham stimulation 10 minutes
- NEMOS device 60 minutes stimulation (Active Comparator): Subjects will be stimulated in the cymba concha with a vibro-tactile mechanical device for 60 minutes
  Interventions: Device: Stimulation 10 minutes; Device: NEMOS transvagal stimulation 60 minutes; Device: NEMOS Device sham stimulation 10 minutes
- Sham 10 minutes (Sham Comparator): 10 minutes of t-VNS stimulation by rotating the NEMOS ear electrode 180 degrees within the pinna, which will position the electrode on the earlobe
  Interventions: Device: Stimulation 10 minutes; Device: NEMOS transvagal stimulation 60 minutes; Device: NEMOS Device sham stimulation 10 minutes

INTERVENTIONS:
Device: Stimulation 10 minutes — NEMOS transvagal stimuli 10 minutes
Device: NEMOS transvagal stimulation 60 minutes — NEMOS Device stimulation in 60 minutes
Device: NEMOS Device sham stimulation 10 minutes

SUMMARY:
This will be a two-stage study to test whether t-VNS using the NEMOS device can activate the CAP and reduce markers of systemic inflammation. Stage A (healthy volunteers) stage B (patients with Juvenile Idiopathic Arthritis).

Stage A: healthy human volunteers. A randomized, single blind, three-period crossover design comparing the CAP activation effect of 10 minutes (active) versus 60 minutes (active) versus 10 minutes (sham) stimulation with the NEMOS device. CAP activation will be assessed by reduction in the in vitro release of LPS-inducible cytokines from whole blood.

Analysis of the reduction in whole blood cytokine release assay after 10 versus 60 minutes of stimulation, and the kinetics of the nadir of the whole blood cytokine release assay will inform the selection of dose duration and sampling time for Stage B. Performing this more extensive exploration of dose duration and kinetics in adults will allow one dose, and a single optimal sampling time in the JIA patients, thus minimizing blood drawing and discomfort in these children.

Stage B will be performed in patients with JIA. This will be an open label design examining the effect of the optimal dose duration (either 10 minutes or 60 minutes of stimulation, as determined by results of Stage A). All information regarding Stage B will be registered in a separate registration at clincialtrials.gov. in order to keep accuracy. All details below concerns only Stage A.

DETAILED DESCRIPTION:
The vagus nerve mediates the "inflammatory reflex"; a mechanism the central nervous system utilizes to regulate innate and adaptive immunity (Andersson, 2012). The afferent arm of the reflex senses inflammation both peripherally and in the central nervous system, and down-regulates the inflammation via efferent neural outflow. The efferent arm of this reflex has been termed the "cholinergic anti-inflammatory pathway" (CAP). The reflex serves as a physiological regulator of inflammation by responding to environmental injury and pathogens with an appropriate degree of immune system activation An increasing body of evidence indicates that the CAP can also be harnessed to reduce pathological inflammation. Electrical neurostimulation of the vagus nerve (VNS) with either a surgically implantable device, or alternatively using a non-invasive device that stimulates the auricular branch of the vagus nerve (ABVN) may be a feasible means of modulating diseases characterized by excessive and dysregulated inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Males and females ages 18-75, inclusive
* Subjects must be free from any active disease, and must not be on any medication that, in the opinion of the investigator, might compromise the measurement or interpretation of the study biomarkers
* Subjects must be able to attend all study visits

Exclusion criteria:

* Significant psychiatric disease or substance abuse
* Anatomic abnormalities, wounds, significant scars or skin disorders affecting the left pinna or external ear canal which would hinder the safe and proper use of the study device
* History of unilateral or bilateral vagotomy
* History of recurrent vasovagal syncope episodes
* Women who are pregnant or plan to conceive during the study. Women of childbearing potential must be willing to use a reliable form of birth control during the study.
* Known history of cardiac rhythm disturbances, atrioventricular block of greater than first degree, or cardiac conduction pathway abnormalities other than isolated right bundle branch block or isolated left anterior fascicle block
* Presence of previously implanted electrically active medical devices (e.g., cardiac pacemakers, automatic implantable cardioverter-defibrillators), or plans to implant such devices during the course of the study
* Planned use of any other external electrically active medical device during the course of the study (e.g., transcutaneous electrical nerve stimulation [TENS] units)
* Any investigational small molecule drug within 30 days of Day 0, visit investigational monoclonal antibody or soluble receptor within 3 months of Day 0 visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Anti-inflammatory Pharmacokinetics | 3 months
  Determine if CAP can be evoked and set the maximum percent change in the in vitro release of LPS-inducible TNF in the whole blood in vitro LPS-inducible cytokine release assay, over the interval from pre-t-VNS to 7 days following t-VNS, comparing sham treatment to each of the two active treatment groups, i.e. 10 minutes and 60 minutes

SECONDARY OUTCOMES:
Anti-inflammatory response | 3 months
  Determine whether 60 minutes of t-VNS induces greater reduction and/or longer duration of effect than 10 minutes as assessed by the in vitro release of LPS-inducible TNF from whole blood
Anti inflammatory response | 3 months
  -Determine the optimum time point for blood sampling the in vitro release of LPS-inducible TNF from whole blood as assessed by the time of nadir post-stimulation
Anti-inflammatory response | 3 months
  Determine the effect of t-VNS on the in vitro release of LPS-inducible IL-1 and IL-6 from whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Andersson, Professor, Study Chair — Department of Women´s and Children´s Health | Karolinska Institutet
Locations (2):
- Sweden (2):
  - Astrid Lindgrens Childrens Hospital, Karolinska University Hospital,, Stockholm, Solna
  - Astrid Lindgren University Hospital, Stockholm, Stockholm County